CLINICAL TRIAL: NCT04668326
Title: Impact of Mobile Manual Standing Wheelchair on Standing Dosage and Utility
Brief Title: Mobile Manual Standing Wheelchair for SCI
Acronym: MMSW-SCI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: F3505-R
Record Dates: First submitted 2020-11-27; First posted 2020-12-16 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injuries and Disorders
Keywords: Paraplegia; Mobility; Standing; Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries; Disease; Paraplegia

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Device Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Manual Standing Wheelchair (Active Comparator): Mobile in seated position; Not mobile in standing position
  Interventions: Device: Manual Standing Wheelchair
- Mobile Manual Standing Wheelchair (Experimental): Mobile in BOTH seated and standing positions
  Interventions: Device: Mobile Manual Standing Wheelchair

INTERVENTIONS:
Device: Manual Standing Wheelchair — Mobile in seated position; Not mobile in standing position
  Other Names: Levo Summit Wheelchair
  Arms: Manual Standing Wheelchair
Device: Mobile Manual Standing Wheelchair — Mobile in BOTH seated and standing positions
  Other Names: Modified Levo Summit Wheelchair
  Arms: Mobile Manual Standing Wheelchair

SUMMARY:
People with spinal cord injuries (SCI) are particularly prone to complications from excessive sitting, because many are not able to stand without support. Excessive sitting after SCI is believed to contribute to pressure injuries, pain, osteoporosis, joint stiffness, spasticity, and worsening bowel and bladder function. The VA has developed, patented, and licensed a mobile manual standing wheelchair (MMSW), and the investigators believe the key feature of being able to wheel around while in a standing position will dramatically change how paralyzed Veterans function in their home and community. If this expanded utility is realized, persons with SCI may naturally spend more time standing and less time sitting. To test these ideas, Veterans with SCI will be randomized to using one of two manual standing wheelchairs at home and in the community for two months.

DETAILED DESCRIPTION:
Background - The investigators contend that for Veterans with SCI to stand enough to impact health outcomes, the standing device must enhance utility while integrating into their everyday life; at home, at work, and in the community. For this integration to occur, the investigators believe the standing device must fulfill the following criteria: 1. Easy access, 2. Straightforward standing mechanism, 3. Mobility in both seated and standing positions, 4. Natural intuitive propulsion, 5. Stability, and 6. Independent operability. The Minneapolis Adaptive Design & Engineering (MADE) Program has recently developed a mobile manual standing wheelchair (MMSW) with all these features. Based on initial in-lab pilot testing, Veterans who trialed the device demonstrated excellent functional mobility and stability in both seated and standing postures. User feedback received during this initial testing also indicated these unique mobility and stability features offer potential new utility for Veterans with SCI.

Research Questions (Objectives) - The purpose of this project is to extend testing of the MMSW to home and community environments of 48 Veterans with SCI to see if mobility in standing affects utility and standing time.

Relevance to VA - There is a mounting body of literature showing significant adverse health consequences associated with excessive time spent in a seated position. Any person who has an underlying condition which impairs their ability to stand or walk is at increased risk for seating related adverse health consequences. There are an estimated 1.7 million people in the United States who have enough impairment that they use seated mobility devices (wheelchairs and scooters). Specifically, people with spinal cord injuries (SCI) are particularly prone to complications from excessive sitting, because many are unable to stand without some type of support. According to the VA's Corporate Data Warehouse, the VA provides care to 17,886 Veterans with SCI/D each year and estimate that over 7,000 of these Veterans have paraplegia. Excessive sitting after SCI is believed to contribute to pressure injuries, worsening pain, osteoporosis, joint stiffness, spasticity, and worsening bowel and bladder function. Until recently, there have been few practical options for safely supporting these individuals while standing or walking. Although there is now a growing list of assistive devices available to support standing and walking in SCI, relatively little attention has been given to determining how often such devices are used or how often they would need to be used to optimally promote the various potential health-related outcomes, nor which devices are most likely to achieve these changes.

Number of Research Participants (Sample Size) - Forty-eight participants (24/group) will be randomized. Each of the two study sites will be expected to screen up to 390 participants to reach the target of 48 randomized over both sites.

Participating Sites - Minneapolis VA Health Care System, VA Palo Alto Health Care System

Duration of Participant Intake (Study Duration) - This project is projected to be a total of four years. The two study sites will have a start-up period of between three to six months and will recruit for approximately three years. The remaining six to nine months will be used for dissemination of study results and study close-out.

Treatment (follow-up) - The intervention being tested is two months of home and community use of a manual standing wheelchair (mobile or non-mobile in standing).

Endpoints - The primary outcomes for this study are utility and standing dose.

Utility - The utility of the study wheelchairs and the current standing device (when applicable) will be assessed using the Wheelchair Outcome Measure (WhOM). The WhOM focuses on ICF constructs of participation and body function. It will be slightly modified to ask users to provide participation goals in the home and community in the context of standing devices/wheelchairs as opposed to wheelchairs alone. The WhOM collects activities that are goals for participation and then has the participant rank the importance and satisfaction with each activity. These rankings allow a quantitative score to be calculated for comparison.

Standing dose - Acceleration data from data loggers will be downloaded and placed on a secure server for further analysis. These data will be visually inspected to determine a threshold for distinguishing sitting and standing postures. These values may vary depending on the mounting on each standing device. After mounting with each system, the participant will go through a sit-to-stand movement and data will be uploaded to ensure the system is detecting movement. This initial movement will also be used to determine an appropriate threshold for standing/sitting. In addition to overall standing time, the investigators will examine frequency of standing bouts and time per standing bout as these are relevant for future pressure injury prevention. The investigators will also monitor movement of the wheelchair during both sitting and standing to understand how often the mobility feature of the MMSW is used during the study.

ELIGIBILITY:
Inclusion Criteria:

* United States Veteran
* SCI or stable disorder/dysfunction of the spinal cord
* Tolerates manual wheelchair use on a regular basis
* Sufficient hand & arm function to operate manual standing wheelchair
* Unable to stand independently without support
* Greater than 6 months post-injury (SCI), or 6 months post diagnosis (disorder/dysfunction)
* Weight less than 125 kg (275 lbs)
* Age 18 or older
* Decisional competency to provide consent and cognitive ability to participate fully in study procedures
* Body size appropriate to fit the devices
* Not involved in another study related to mobility
* Identify an appropriate location for use of the study wheelchair

Exclusion Criteria:

* Contraindication for standing including lower limb contractures, uncontrolled hypertension, uncontrolled spasticity, etc.
* Unhealed lower-limb fractures
* Unstable lower-limb joints
* An active grade 2 or greater pressure injury that can be worsened by standing in the device
* Flap procedure to address pressure injury less than one year earlier
* Not able to propel a manual wheelchair or operate the sit-to-stand mechanism (e.g. weakness, or discomfort)
* Low bone mineral density (BMD), defined by total hip DXA more than 3.5 SD below peak and/or distal femur/proximal tibia BMD below 0.6 g/cm2. (Low BMD at any site will be ineligible).
* Unable to obtain clinically acceptable seating system for study wheelchairs
* Unable to build up standing tolerance within the first eight visits
* Individual deemed not appropriate for participation in the study as determined by study team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Utility - Measured using the Wheelchair Outcome Measure | Two months
  The Wheelchair Outcome Measure (WhOM) will be slightly modified to ask users to provide participation goals in the home and community in the context of standing devices/wheelchairs as opposed to wheelchairs alone. The WhOM collects activities that are goals for participation and then has the participant rank the importance and satisfaction with each activity. The rankings allow a quantitative score to be calculated for comparison. The WhOM was chosen to represent the concept of "utility" because it captures what is meaningful and important to each participant, while also allowing a quantitative scoring.
  The investigators will specifically calculate Mean satisfaction x importance = the sum of the individual importance x satisfaction of all goals divided number of goals
  Higher scores indicate higher satisfaction with specific goals, using importance of the task to help scale the effect of each goal. Thus higher scores will be considered higher utility.
Standing Dose - Total time standing - Study Wheelchair | Two months
  An accelerometer will be placed on part of the study standing wheelchair that rotates upward during standing. The gravitational acceleration will indicate standing versus sitting. A custom algorithm will be used to determine when the wheelchair is in the standing position.
Standing Dose - Total time standing - Existing Standing Device | Two months
  An accelerometer will be placed on part of the existing standing device (when applicable) that rotates upward during standing. The gravitational acceleration will indicate standing versus sitting. A custom algorithm will be used to determine when the standing device is in the standing position.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew H Hansen, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN; B. Jenny Kiratli, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (2):
- United States (2):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-07-24): https://cdn.clinicaltrials.gov/large-docs/26/NCT04668326/ICF_000.pdf